CLINICAL TRIAL: NCT00972348
Title: A Randomized Controlled Trial Embedded in an Electronic Medical Record (myHERO).
Brief Title: Trial Embedded in an Electronic Personal Medical Health Records
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H2598-33964; R18HS017784 (AHRQ)
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections; Health Literacy
Keywords: HIV; Personal Health Record; Laboratory values: CD4 cells and HIV Viral load; Medication Reconciliation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Access to Personal Health Record (Experimental): Full access to the Personal Health Record including lists of diagnoses, medications and laboratory values.
  Interventions: Other: Online access to a personal health record
- No access to the PHR (Active Comparator): No access to the PHR but patients will complete surveys.
  Interventions: Other: No access to the PHR

INTERVENTIONS:
Other: Online access to a personal health record — Patients in the intervention arm have full access to their online personal health record
  Arms: Access to Personal Health Record
Other: No access to the PHR — Patients will not be given access to their PHR but will complete online surveys.
  Arms: No access to the PHR

SUMMARY:
This is a research study to determine if a personal health record, called myHERO, will help improve health. A personal health record is a secure internet (also called online) tool that contains personal health information like medications, diagnosed conditions, allergies and laboratory values (like CD4 cells and viral load). This study will also help explain if a personal health record influences the relationship with a doctor or nurse practitioner and their patients. The purpose of this study is to determine if a personal health record will influence health. The content of your personal health record is as secure as possible for any online health information.

DETAILED DESCRIPTION:
HIV/AIDS is a non-curable chronic illness. Applying the chronic care model (CCM) to this disease may lead to improved outpatient based health care and easier clinical transitions for HIV infected patients. Clinical information systems (CIS) are a key element in the CCM and have three important roles: reminder systems; feedback mechanisms; and registries. CIS have focused on the provider as the recipient of critical data, however clinical information systems that target patients as consumers of information might also contribute to improved health care, especially for ambulatory patients. Personal health records (PHRs) are tools that would fit as a clinical information system for patients. PHRs allow patients (and others) to view data that are necessary to guide practical outpatient decisions. PHRs can become platforms to support the CIS elements too, allowing patients to receive and understand information, engage in their healthcare and influence their health outcomes. Our central hypothesis is that a secure enhanced PHR (ePHR) that combines meaningful information, web-based tools for support and reminders for patients will also provide a substantial opportunity to promote self-management and will lead to improved health outcomes. In this proposal we will work directly with HIV/AIDS patients in a public health setting to model processes that contribute to improved health outcomes in the realms of patient behaviors, patient-clinician trust, clinical outcomes, medication safety and utilization. Accordingly, the specific aims are:

1. (Build Infrastructure and Content) Extend and secure a web-based PHR for HIV/AIDS patients receiving care in a public health setting providing these users with tools to access and understand their medical record including resources for decision support, information retrieval and communication. Specific content will include access to support for tobacco cessation, depression abatement, anxiety reduction, and medication adherence improvement.
2. (Evaluation of PHR) Evaluation of patient and clinician experience with PHR including patient access and use patterns including use of support for tobacco cessation, depression abatement, anxiety reduction, adherence improvement., patient and clinician satisfaction with ePHR.
3. (Outcome Assessment) Evaluation in 5 domains: quality of the patient-clinician interaction (trust, communication, health promotion); changes in patient behaviors (risk behaviors, adherence to antiretroviral medications, tobacco use); clinical outcomes (CD4+ T-lymphocytes, detectable plasma HIV RNA, depression, anxiety, quality of life); safety (documentation of drug allergies, adverse events, medication reconciliation); and utilization (office visits).

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of HIV-1 infection, based on patient's medical history or laboratory tests.
2. 18 years of age or older
3. Receiving primary medical care at the Positive Health Program, SFGH.
4. Able and willing to give informed consent.
5. Willing to use the patient portal

Exclusion Criteria:

1. Unwilling or unable to provide informed consent.
2. No access to the web at any convenient location.
3. Not willing to respond to online surveys or questionnaires.
4. Already with access to the myHERO system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary analyses of the trial data will compare the two study groups with respect to (1) 12-month change in CD4 T-cell count and (2) 12-month proportion of patients whose HIV viral load (VL) level is detectable. | 12 months of participation

SECONDARY OUTCOMES:
Alleviation of depression, among patients who are depressed at baseline. | 12 months
Smoking cessation, among patients who are smokers at baseline. | 12 months
Trust between physicians and patients. | 12 months
Medication reconciliation. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James Kahn, MD, Principal Investigator — University of California; David Thom, MD, PhD, Study Director — University of California, San Francisco
Locations (1):
- HIV AIDS outpatient clinic at Ward 86, San Francisco, California, United States